CLINICAL TRIAL: NCT04123145
Title: Study of the Prevalence of Iron Deficiency in Patients With Chronic Renal Failure But Non-Dialysis (CARENFER IRC-ND)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VIFORFRANCE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CARENFER IRC
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDK-ND (Experimental)
  Interventions: Diagnostic Test: Iron status testing

INTERVENTIONS:
Diagnostic Test: Iron status testing — Iron status testing

SUMMARY:
Despite its known prevalence, a recent study conducted with Prof. Cacoub (unpublished) on the national health insurance database showed that iron deficiency was a poorly diagnosed and poorly treated comorbidity. In patients with Chronic Kidney Disease but Non-Dialysis, the determination of Ferritinemia and Transferrin Saturation Factoris performed in only 30% and 10% of cases whereas they should be performed routinely in inflammatory situations and in case of anemia (HAS 2011, KDIGO 2012). The objective of this study is to obtain updated data on the prevalence of iron deficiency in France in patients with CKD-ND, applying the international recommendations and those of the French Health High Authority (determination of ferritinemia and Transferrin Saturation Factor).

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years of age;
* Patient present at the hospital on the day of the study (traditional hospitalization, week hospital, day hospital, or in consultation with CKD-ND);
* Diagnosis of CKD-ND (glomerular filtration rate (GFR) > 15 mL/min/1.73 m²)
* Patient with signed consent

Exclusion Criteria:

* Protected patient: major under guardianship, tutorship or other legal protection, deprived of liberty by judicial or administrative decision;
* Pregnant or breastfeeding woman;
* Patient with dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2019-10-15 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Complete blood iron status | One day
  ferritin
Complete blood iron status | One day
  Transferrin Saturation Factor

IPD SHARING:
Plan to Share IPD: No